CLINICAL TRIAL: NCT07071441
Title: Rectal Indomethacin Versus Diclofenac for Prevention of Post-ERCP Panceratitis (IDPPP2): A Multicenter, Double-blind, Randomized, Control Trial
Brief Title: Indomethacin vs Diclofenac for Preventing PEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20242439-F-1
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: ERCP; Pancreatitis; Non-steroidal Anti-inflammatory (NSAID); Indomethacin; Diclofenac
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indomethacin (Experimental): All patients without contraindications should receive 100mg rectal indomethacin within 30mins before ERCP procedure
  Interventions: Drug: Indomethacin 100 MG
- Diclofenac group (Active Comparator): All patients without contraindications should receive 100mg rectal diclofenac within 30mins before ERCP procedure
  Interventions: Drug: Diclofenac 100mg

INTERVENTIONS:
Drug: Indomethacin 100 MG — All patients without contraindications should receive 100mg rectal indomethacin within 30mins before ERCP procedure
  Arms: Indomethacin
Drug: Diclofenac 100mg — All patients without contraindications should receive 100mg rectal diclofenac within 30mins before ERCP procedure
  Arms: Diclofenac group

SUMMARY:
Pancreatitis is the most common and serious complication following post-endoscopic retrograde cholangiopancreatography (ERCP) and is associated with occasional mortality, extended hospital stays, and increased healthcare expenses. Preprocedural administration of rectal non-steroidal anti-inflammatory drugs (NSAIDs) was demonstrated to be an effective and convenient strategy for post-ERCP pancreatitis (PEP). Furthermore, several meta-analyses found that only 100mg indomethacin and diclofenac could effectively reduce PEP. Therefore, updated international clinical practice guidelines uniformly recommended administration of 100mg indomethacin or diclofenac in patients without contradictions. However, it was unclear which one of the two drug is more superior.

A recent meta-analysis suggested 100mg rectal diclofenac was more efficacious than same-dose rectal indomethacin in PEP prevention (relative risk (RR) 0·59, 95% confidence intervals (CI) 0·40-0·89). Based on the results, we conducted a multicenter, double-blind, control trial to investigate whether 100mg diclofenac is superior than same-dose indomethacin. This trial planned to enroll 3612 patients in total. However, in the first interim analysis, PEP occurred in 53 patients (8.8%) of 600 patients allocated to diclofenac group and 37 patients (6.1%) of 604 patients allocated to indomethacin group (relative risk (RR) 1.44; 95% confidence interval (CI) 0.96-2.16, p=0.074). Thus, the trial was stopped according to the futility rule of conditional power. However, it was worth noticing that PEP tended to be higher in diclofenac group than that in indomethacin group. A sample size of 1204 was under power to draw the conclusion of significantly lower PEP rate in indomethacin group and thus a new trial with larger sample size of sufficient power is predicted to prove the superiority of indomethacin over diclofenac. Here we conducted a multicenter, randomized, double-blind trial to investigate whether 100mg indomethacin is superior to 100mg diclofenac in preventing PEP.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old patients with native papilla who planned to undergo ERCP

Exclusion Criteria:

* Previous biliary sphincterotomy and papillary large balloon dilation
* Planned for placements of pancreatic duct stents (eg. pancreatic duct strictures, planned ampullectomy)
* Allergy to NSAIDs
* The administration of NSAIDs within 7 days
* Not suitable for NSAIDs administration (gastrointestinal hemorrhage within 4 weeks, renal dysfunction [Cr >1.4mg/dl=120umol/l]; presence of coagulopathy before the procedure)
* Acute pancreatitis within 7 days before ERCP or acute pancreatitis with obvious Pancreatic edema and peripancreatic fluid collections
* Hemodynamical instability
* Pregnancy or lactation
* Unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4050 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of post-ERCP Pancreatitis | 30 days
  a new or aggravated upper abdominal pain, with an elevated pancreatic enzyme of at least 3 times as the upper limit of normal value 24h after procedure and prolonged hospitalization days for at least 2 days. This definition was based on a widely recognized Cotton consensus

SECONDARY OUTCOMES:
Rate of mild, moderate or severe PEP | 30 days
  The severity classification of post-ERCP pancreatitis was defined according to the Cotton Criteria. Mild PEP: with an extension of hospitalization period of 2-3 days; Moderate PEP: with an extension of hospitalization period of 4-10 days; Severe PEP: with an extension of more than 10 days, or hemorrhagic pancreatitis, phlegmon, or pseudocyst, intervention (percutaneous drainage or surgery), or death.
Rate of patients with different severity of pancreatitis evaluated by revised Atlanta criteria | 30 days
  Mild: The most common form of acute pancreatitis, without organ failure or local or systemic complications, generally resolving within 1 week of onset.
  Moderately Severe: the presence of transient organ failure, local complications or exacerbation of co-morbid disease.
  Severe: persistent organ failure, that is, organ failure >48 h. Local complications are peripancreatic fluid collections, pancreatic and peripancreatic necrosis (sterile or infected), pseudocyst and walled-off necrosis (sterile or infected).
Rate of ERCP-related perforation | 30 days
  Perforation was established according to Cotton criteria, Mild: slight leakage of fluid or contrast dye, manageable through fluid administration and suction therapy ≤3 days Moderate: definite perforation required to be managed for 4-10 days Severe: management for more than 10 days or requiring for percutaneous or surgical intervention.
Rate of ERCP-related infection | 30 days
  Infection was established according to Cotton criteria. Mild: temperature >38℃ for 24-48h Moderate: Febrile illness requiring >3 days of hospital treatment; endoscopic or percutaneous interventions; Severe: septic shock or requiring surgery.
Rate of ERCP-related bleeding | 30 days
  Bleeding was established according to Cotton criteria. Mild: a documented decrease in hemoglobin concentration by <3 g/L, without requiring the blood transfusion; Moderate: blood transfusion ≤4 units; without need for angiographic or surgery interventions Severe: Transfusion: ≥5 units or requiring for angiographic or surgery interventions.
Rate of NSAIDs-related complications | 30 days
  NSAIDs-related complications include: acute kidney injury, allergic reaction, gastrointestinal bleeding, myocardial infarction, cerebrovascular accident, and death
Rate of mortality | 30 days
The rate of total adverse events | 30 days
  Adverse events include ERCP-related or non ERCP-related adverse events

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - The first medical center, Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Department of Gastroenterology, Hongai Hospital, Xiamen, Fujian
  - Harbin Medical University Affiliated Fourth Hospital, Harbin, Heilongjiang
  - Zhaolei181220@163.Com, Harbin, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Hennan
  - Renmin hospital of Wuhan University, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jilin Miniciple People'S Hospital, Jilin, Jilin
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - 986 Hospital of Xijing Hospital, Xi'an, Shaanxi
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - The 960th Hospital of the PLA, Jinan, Shandong
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - the second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akshintala VS, Sperna Weiland CJ, Bhullar FA, Kamal A, Kanthasamy K, Kuo A, Tomasetti C, Gurakar M, Drenth JPH, Yadav D, Elmunzer BJ, Reddy DN, Goenka MK, Kochhar R, Kalloo AN, Khashab MA, van Geenen EJM, Singh VK. Non-steroidal anti-inflammatory drugs, intravenous fluids, pancreatic stents, or their combinations for the prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis: a systematic review and network meta-analysis. Lancet Gastroenterol Hepatol. 2021 Sep;6(9):733-742. doi: 10.1016/S2468-1253(21)00170-9. Epub 2021 Jun 30. PMID 34214449
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Kang X, Xia M, Wang J, Wang X, Luo H, Qin W, Liang Z, Zhao G, Yang L, Sun H, Tao J, Ning B, Zhong L, Zhang R, Ma X, Zhao J, Yue L, Jin H, Kang C, Ren G, Liang S, Wang H, Wang L, Nie Y, Wu K, Fan DM, Pan Y. Rectal diclofenac versus indomethacin for prevention of post-ERCP pancreatitis (DIPPP): a multicentre, double-blind, randomised, controlled trial. Gut. 2025 Jun 6;74(7):1094-1102. doi: 10.1136/gutjnl-2024-334466. PMID 40113243
- [Background] Luo H, Zhao L, Leung J, Zhang R, Liu Z, Wang X, Wang B, Nie Z, Lei T, Li X, Zhou W, Zhang L, Wang Q, Li M, Zhou Y, Liu Q, Sun H, Wang Z, Liang S, Guo X, Tao Q, Wu K, Pan Y, Guo X, Fan D. Routine pre-procedural rectal indometacin versus selective post-procedural rectal indometacin to prevent pancreatitis in patients undergoing endoscopic retrograde cholangiopancreatography: a multicentre, single-blinded, randomised controlled trial. Lancet. 2016 Jun 4;387(10035):2293-2301. doi: 10.1016/S0140-6736(16)30310-5. Epub 2016 Apr 28. PMID 27133971